CLINICAL TRIAL: NCT06039306
Title: Perioperative Immunonutrition Among Gynecological Cancer Patients Under Enhanced Recovery After Surgery
Brief Title: Perioperative Immunonutrition Under Enhanced Recovery After Surgery
Acronym: PING-ERAS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, ChiouYi Ho, Principal Investigator, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RSCH ID-22-04215-WHE
Record Dates: First submitted 2023-08-24; First posted 2023-09-15 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2024-08

CONDITIONS: Gynecological Cancer; Elective Surgery
Keywords: gynecological cancer, elective surgery

STUDY DESIGN:
Intervention Model Description: After consented, participants will be randomized into two groups: the intervention group and conventional group during consultation in multidisciplinary clinic.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): Participants will be given 2 servings immunonutrition daily for five (5) days before tentative elective surgery. ERAS protocol will implement and continued 2 servings of immunonutrition for post-operative seven (7) days.
  Interventions: Dietary Supplement: Immunonutrition oral nutrition supplementation
- conventional (No Intervention): Participants will be on usual diet intake before tentative elective surgery. ERAS protocol will implement and will be prescribed 2 servings of polymeric formula daily only if unable to finish 75% of the diet served in ward.

INTERVENTIONS:
Dietary Supplement: Immunonutrition oral nutrition supplementation — Participant will prescribed with 2 servings of immunonutrition supplement 5 days before surgery and 7 days after surgery
  Arms: intervention

SUMMARY:
The goal of this clinical trial is to compare the effect of perioperative immunonutrition supplement in gynecologic cancer patients. The main questions it aims to answer are:

* is there any difference in the nutritional outcomes and functional outcomes between intervention and conventional groups?
* is there any difference in the post-surgical outcomes between intervention and conventional groups?

Participants (intervention) will be provided the immunonutrition supplement before and after operation.

Researchers will compare intervention group with conventional group to see if there is any difference in postoperative outcomes.

DETAILED DESCRIPTION:
The clinical trial aims to determine the effectiveness of perioperative IMN intervention on postoperative outcomes among GC patients under Enhanced Recovery after Surgery (ERAS) setting. Patients will prescribed with immunonutrition supplement before and after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Those who diagnosed with GC
2. Candidates for elective operation treatments

Exclusion Criteria:

1. Those are involved gastrointestinal tract (complication)
2. Those are diagnosed with GC (metastasis)
3. Allergy to milk/soy/whey protein
4. Participate in other intervention study

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
daily energy and protein intake | 1 month
  24-hours diet recall
body composition | 1 month
  body composition analyzer; weight in kg; fat free mass in kg; fat mass in kg; muscle mass in kg; height in meter
immunoglobulin level | 1 month
  Concentration of immunoglobulin G; Concentration of immunoglobulin A; Concentration of immunoglobulin M
C-reactive protein | 1 month
  Concentration of C-reactive protein
postoperative outcomes | 1 months
  length of hospitalization

SECONDARY OUTCOMES:
Functional status | 1 month
  handgrip strength in kg via Jammar dynamometer
stress level | 1 month
  questionnaire 10-item perceived stress scale (PSS-10) form

CONTACTS AND LOCATIONS:
Overall Officials: ChiouYi Ho, Principal Investigator — National Cancer Institute, Malaysia
Locations (1):
- Institut Kanser Negara, Putrajaya, Putrajaya, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hertlein L, Zeder-Goss C, Furst S, Bayer D, Trillsch F, Czogalla B, Mahner S, Burges A, Rittler P. Peri-operative oral immunonutrition in malnourished ovarian cancer patients assessed by the nutritional risk screening. Arch Gynecol Obstet. 2018 Jun;297(6):1533-1538. doi: 10.1007/s00404-018-4759-8. Epub 2018 Apr 5. PMID 29623417
- [Background] Abeles A, Kwasnicki RM, Darzi A. Enhanced recovery after surgery: Current research insights and future direction. World J Gastrointest Surg. 2017 Feb 27;9(2):37-45. doi: 10.4240/wjgs.v9.i2.37. PMID 28289508
- [Background] Arends J, Bachmann P, Baracos V, Barthelemy N, Bertz H, Bozzetti F, Fearon K, Hutterer E, Isenring E, Kaasa S, Krznaric Z, Laird B, Larsson M, Laviano A, Muhlebach S, Muscaritoli M, Oldervoll L, Ravasco P, Solheim T, Strasser F, de van der Schueren M, Preiser JC. ESPEN guidelines on nutrition in cancer patients. Clin Nutr. 2017 Feb;36(1):11-48. doi: 10.1016/j.clnu.2016.07.015. Epub 2016 Aug 6. PMID 27637832
- [Background] Ho CY, Ibrahim Z, Abu Zaid Z, Mat Daud ZA, Mohd Yusop NB, Mohd Abas MN, Omar J. Postoperative Dietary Intake Achievement: A Secondary Analysis of a Randomized Controlled Trial. Nutrients. 2022 Jan 5;14(1):222. doi: 10.3390/nu14010222. PMID 35011097
- [Background] Yi HC, Ibrahim Z, Abu Zaid Z, Mat Daud Z', Md Yusop NB, Omar J, Mohd Abas MN, Abdul Rahman Z, Jamhuri N. Impact of Enhanced Recovery after Surgery with Preoperative Whey Protein-Infused Carbohydrate Loading and Postoperative Early Oral Feeding among Surgical Gynecologic Cancer Patients: An Open-Labelled Randomized Controlled Trial. Nutrients. 2020 Jan 20;12(1):264. doi: 10.3390/nu12010264. PMID 31968595
- [Background] Mudge LA, Watson DI, Smithers BM, Isenring EA, Smith L, Jamieson GG; Australian Immunonutrition Study Group. Multicentre factorial randomized clinical trial of perioperative immunonutrition versus standard nutrition for patients undergoing surgical resection of oesophageal cancer. Br J Surg. 2018 Sep;105(10):1262-1272. doi: 10.1002/bjs.10923. Epub 2018 Jul 12. PMID 29999517
- [Background] Di Renzo L, De Lorenzo A, Fontanari M, Gualtieri P, Monsignore D, Schifano G, Alfano V, Marchetti M; SIERR. Immunonutrients involved in the regulation of the inflammatory and oxidative processes: implication for gamete competence. J Assist Reprod Genet. 2022 Apr;39(4):817-846. doi: 10.1007/s10815-022-02472-6. Epub 2022 Mar 30. PMID 35353297
- [Derived] Ho C, Daud ZAM, Mohd Yusof BN, Abdul Majid H. Perioperative immunonutrition intervention on postoperative outcomes among gynecological cancer patients under enhanced recovery after surgery setting: A study protocol of explanatory mixed method study. PLoS One. 2024 Dec 31;19(12):e0315568. doi: 10.1371/journal.pone.0315568. eCollection 2024. PMID 39739975